CLINICAL TRIAL: NCT00212420
Title: Nutritional Management of Acute and Chronic Enterocutaneous Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: St Mark's Hospital Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/Q0405/CEF106
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Enterocutaneous Fistulae
Keywords: fistula; enterocutaneous; nutrition;enteral; parenteral; TPN
MeSH Terms: conditions — Fistula | interventions — Parenteral Nutrition; Enteral Nutrition

INTERVENTIONS:
Procedure: parenteral nutrition; enteral nutrition

SUMMARY:
To Investigate whether different routes of nutrition affect the probability of fistula closure in patients with an enterocutaneous fistula

DETAILED DESCRIPTION:
Enterocutaneous fistulae are abnormal connections between bowel and skin through which bowel contents pass. Their management present a considerable medical and surgical challenge. Since the 1970s the mainstray of treatment has been supportive with initiation of a "nil by mouth" regimen and intravenous (parenteral) nutrition with the aim of stabilising the patient and inducing gastrointestinal tract rest. There seems to have been an unquestioned benefit attributed to total parenteral nutrition (TPN) in the 1970s and 1980s which has carried through to the current day. This rigid approach to the management of enterocutaneous fistulae is almost universal and yet an extensive literature search suggests both mixed results from clinical trials and mixed opinions from experts in the field.

A large study published in the late 1970s (Souters et al. 1979) demonstrated that there was a 44% mortality in patients with an enterocutaneous fistula from 1946 to 1959 which fell to 15% between 1960 and 1970 with the introduction of improved parasurgical care; after 1970 no further decrease in mortality rate was observed despite the introduction of parenteral nutrition. It could therefore be argued that parenteral nutrition offers no real additional benefit to these patients. Surprisingly there is no information in the literature comparing enteral nutrition with parenteral nutrition in patients with an enterocutaneous fistula.

Enter nutrition is more physiological, is associated with fewer complications and is cheaper when compared to parenteral nutrition. If parenteral nutrition were shown to offer no benefit with regards to fistula closure in patients with enterocutaneous fistula then enteral feeding would be the nutritional modality of choice. This would constitute a major shift in the current management of such patients.

Recent research has shown that the supply of nutrients to the lining of the gastrointestinal tract can have a significant effect on the growth of the cells lining the gut and on the motility as a whole. Many of these effects are mediated by intestinal growth factors such and glucagon-like peptide-2 (GLP-2) and gut hormones such as cholecystokinin (CCK) and peptide YY (YYY. Although no studies have been performed looking at the levels of growth factors and gut hormones in patients with enterocutaneous fistulae, it seems theoretically likely that the route of nutrition in these patients will have an effect on the levels of these intestinal growth factors and gut hormones. This in turn may have effect on fistula healing and fistula output. Modulation of the levels of these growth factors and gut hormones may provide new therapeutic options in the future management of enterocutaneous fistulae.

ELIGIBILITY:
Inclusion Criteria:

* patients with an enterocutaneous fistula for > 14 days who have been referred to the Nutrition Team (or Pharmacy) for initiation of parenteral nutrition

Exclusion Criteria:

* generalised peritonitis or systemic sepsis (SIRS)
* immediate need for surgery or radiological drainage procedures
* other contraindicators to either enteral or parenteral feeding
* age < 18 years old
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-12

PRIMARY OUTCOMES:
To investigate whether different routes of nutrition affect the probability of fistula closure in patients with an enterocutanous fistula

SECONDARY OUTCOMES:
investigating if different routes of nutrition affect fistula output, complication rates, overall nutrition and quality of life in patients with an enterocutaneous fistula. To measure the levels of intestinal growth factors and gut hormones in patients

CONTACTS AND LOCATIONS:
Overall Officials: David AJ Lloyd, MA, MRCP, Principal Investigator — St Mark's Hospital, North West London NHS Trust
Locations (1):
- St Mark's Hospital, North West London Hospitals NHS Trust, Harrow, Middlesex, United Kingdom